CLINICAL TRIAL: NCT01569113
Title: A Prospective, Randomized, Double-blind Parallel-arm, Placebo-controlled Study to Assess the Effects on Ovarian Activity of a Combined Oral Contraceptive Pill When Preceded by the Intake of ellaOne® (Ulipristal Acetate 30 mg) or Placebo.
Brief Title: Assessment of Effects on Ovarian Activity of a Combined Oral Contraceptive Pill When Preceded by the Intake of ellaOne® or Placebo.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2914-015
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Emergency Contraception
Keywords: ella; ellaOne; quickstart; contraception; combined oral pill; microgynon
MeSH Terms: interventions — ulipristal acetate; Ethinyl Estradiol; Levonorgestrel; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ellaOne + microgynon 30 (Experimental)
  Interventions: Drug: Ulipristal Acetate (UPA) + ethinylestradiol/levonorgestrel (Microgynon)
- placebo + microgynon 30 (Placebo Comparator)
  Interventions: Drug: placebo + ethinylestradiol/levonorgestrel

INTERVENTIONS:
Drug: Ulipristal Acetate (UPA) + ethinylestradiol/levonorgestrel (Microgynon) — UPA: 30 mg, 1 tablet, single intake Microgynon 30mcg/150mcg, 1 tablet per day, 21-day intake
  Other Names: ellaOne + Microgynon 30
  Arms: ellaOne + microgynon 30
Drug: placebo + ethinylestradiol/levonorgestrel — placebo: 1 tablet, single intake Microgynon 30mcg/150mcg, 1 tablet per day, 21-day intake
  Other Names: Microgynon 30
  Arms: placebo + microgynon 30

SUMMARY:
The purposes of this study are to compare the effects on ovarian activity of quick starting a Combined Oral Contraceptive Pill (COCP) after ellaOne® or placebo intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-35 years old
* BMI < 30 Kg/m2
* Not at risk of pregnancy
* No use of progesterone-only-pill for 3 months before start of treatment cycle
* No use of implant hormonal contraception for 3 months before start of treatment cycle
* No use of levonorgestrel intrauterine system for 3 months before start of treatment cycle
* No use of depo provera for 12 months before start of treatment cycle
* Able to give informed consent.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a Hoogland score consistent with ovarian quiescence (≤3) after 1 to 21 days of intake of COCP in both groups (preceded by the intake of ellaOne® or placebo). | Day 1 to day 21 of intake of microgynon 30

SECONDARY OUTCOMES:
Number of days of intake of COCP required to reach ovarian quiescence (Hoogland score ≤3) after the intake of ellaOne® or placebo. | Day 1 to day 21 of intake of microgynon 30

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Cameron, MD, Principal Investigator — Chalmers Sexual Health Clinic
Locations (3):
- Dinox, Groningen, Netherlands
- Karolinska University Hospital Solna, Stockholm, Sweden
- Chalmers Sexual Health Clinic, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Derived] Cameron ST, Berger C, Michie L, Klipping C, Gemzell-Danielsson K. The effects on ovarian activity of ulipristal acetate when 'quickstarting' a combined oral contraceptive pill: a prospective, randomized, double-blind parallel-arm, placebo-controlled study. Hum Reprod. 2015 Jul;30(7):1566-72. doi: 10.1093/humrep/dev115. Epub 2015 May 20. PMID 25994664